CLINICAL TRIAL: NCT04734990
Title: Phase I/II Study of SP-2577 (Seclidemstat) in Combination With Azacitidine for Patients With Myelodysplastic Syndromes and Chronic Myelomonocytic Leukemia
Brief Title: Seclidemstat and Azacitidine for the Treatment of Myelodysplastic Syndrome or Chronic Myelomonocytic Leukemia
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0487; NCI-2020-14163 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0487 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-01-28; First posted 2021-02-02 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Chronic Myelomonocytic Leukemia-0; Chronic Myelomonocytic Leukemia-1; Chronic Myelomonocytic Leukemia-2; Myelodysplastic Syndrome; Recurrent Chronic Myelomonocytic Leukemia; Recurrent Myelodysplastic Syndrome
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic | interventions — Azacitidine; seclidemstat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (azacitidine, seclidemstat) (Experimental): Patients receive azacitidine IV over 10-40 minutes or SC on days 1-7. Patients also receive seclidemstat PO QD on day 1 of cycle 1 and PO BID on days 2-28 of cycle 1 and on days 1-28 of all subsequent cycles. There are 6 planned dose levels for seclidemstat: 300 mg, 450 mg, 600 mg, 900 mg, 1200 mg and 1500 mg. Successive cohorts of eligible patients will be treated with azacitidine. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Azacitidine; Drug: Seclidemstat

INTERVENTIONS:
Drug: Azacitidine — Given IV or SC
  Other Names: 5 AZC; 5-AC; 5-Azacytidine; 5-AZC; Azacytidine; Azacytidine, 5-; Ladakamycin; Mylosar; Onureg; U-18496; Vidaza
Drug: Seclidemstat — Given PO
  Other Names: LSD1 Inhibitor SP-2577; SP 2577; SP-2577; SP2577

SUMMARY:
This phase I/II trial identifies the best dose of seclidemstat when given together with azacitidine in treating patients with myelodysplastic syndrome or chronic myelomonocytic leukemia. Seclidemstat may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Azacitidine may help block the formation of growths that may become cancer. Giving seclidemstat and azacytidine may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety, tolerability and maximum tolerable dose (MTD) of seclidemstat in combination with azacitidine.

II. To assess overall response rate (ORR) to seclidemstat in combination with azacitidine.

SECONDARY OBJECTIVES:

I. To assess overall survival (OS), duration of response (DOR), relapse-free survival (RFS), and leukemia-free survival (LFS) and safety profile.

II. Correlative studies including correlation of response with disease subtypes, genomic profile and in vitro studies.

OUTLINE: This is a phase I, dose-escalation study of seclidemstat followed by a phase II dose-expansion study.

Patients receive azacitidine intravenously (IV) over 10-40 minutes or subcutaneously (SC) on days 1-7. Patients also receive seclidemstat orally (PO) once daily (QD) on day 1 of cycle 1 and PO twice daily (BID) on days 2-28 of cycle 1 and on days 1-28 of all subsequent cycles. There are 6 possbile dose levels for seclidemstat: 300 mg, 450 mg, 600 mg, 900 mg, 1200 mg and 1500 mg. Successive cohorts of eligible patients will be treated with azacitidine until the phase 2 recommended dose or maximum tolerated dose is determined. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days, and then every 6 months thereafter

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years as myelodysplastic syndrome (MDS) is a very rare disease in the pediatric setting
* Diagnosis of MDS or chronic myelomonocytic leukemia (CMML) according to World Health Organization (WHO) and:

  * MDS with int-1, int-2, or high risk by International Prognostic Scoring System (IPSS), or CMML-1/CMML-2 , myeloproliferative CMML (white blood cell [WBC] >= 13 x 10^9/L) or CMML-0 with high-risk molecular features (known mutations in ASXL1, SETBP1, RUNX1, NRAS, TP53 or more than 3 mutations).
  * No response after 6 cycles of azacitidine, decitabine, guadecitabine, ASTX030 or ASTX727 or relapse or progression after any number of cycles
* Serum creatinine =< 1.5 x upper limit of normal (ULN) OR creatinine clearance >= 50 ml/min for patients with creatinine levels > 1.5 x ULN
* Adequate hepatic function with total bilirubin < 2 x ULN (will allow less than 5 x ULN if Gilbert's syndrome at investigator's discretion)
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) =< 3 x ULN
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Patient (or patient's legally authorized representative) must have signed an informed consent document indicating that the patient understands the purpose of and procedures required for the study and is willing to participate in the study
* Prior hydroxyurea for control of leukocytosis or use of hematopoietic growth factors (e.g., granulocyte colony-stimulating factor [G-CSF], granulocyte-macrophage colony-stimulating factor [GM-CSF], Procrit, Aranesp, thrombopoietins) is allowed at any time prior to or during study if considered to be in the best interest of the patient

Exclusion Criteria:

* Uncontrolled infection not adequately responding to appropriate antibiotics
* New York Heart Association (NYHA) class III or IV congestive heart failure or left ventricular ejection fraction (LVEF) < 50% by echocardiogram or multigated acquisition (MUGA) scan
* History of myocardial infarction within the last 6 months or unstable/uncontrolled angina pectoris or history of severe and/or uncontrolled ventricular arrhythmias
* Baseline corrected QT interval by Fridericia formula (QTcF) (Fridericia) >= 450 msecs and long QT syndrome or family history of idiopathic sudden death or congenital long QT syndrome
* Currently receiving any of the following substances and cannot be discontinued 14 days for CYP inhibitors prior to cycle 1 day 1:

  * Moderate or strong inhibitors or inducers of major CYP isoenzymes, including grapefruit, grapefruit hybrids, pomelos, star fruit and Seville oranges
  * Moderate or strong inhibitors or inducers of major drug transporters
  * Substrates of CYP3A4/5 with a narrow therapeutic index
* Female patients who are pregnant or lactating
* Patients with reproductive potential who are unwilling to following contraception requirements (including condom use for males with sexual partners, and for females: prescription oral contraceptives [birth control pills], contraceptive injections, intrauterine devices [IUD], double-barrier method [spermicidal jelly or foam with condoms or diaphragm], contraceptive patch, or surgical sterilization) throughout the study
* Female patients with reproductive potential who do not have a negative urine or blood beta-human chorionic gonadotropin (beta human chorionic gonadotropin [HCG]) pregnancy test at screening
* Patients receiving any other concurrent investigational agent or chemotherapy, radiotherapy, or immunotherapy
* Evidence of graft versus host disease or prior allogeneic (allo)-stem cell transplantation within 6 months of cycle 1 day 1 or receiving immunosuppressants following a stem-cell procedure
* Patients known to be positive for hepatitis B surface antigen expression or with active hepatitis C infection (positive by polymerase chain reaction or on antiviral therapy for hepatitis C within the last 6 months). Patients with history of human immunodeficiency virus (HIV) disease are also excluded from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2021-07-07 (Actual); Primary Completion 2027-09-11 (Estimated); Study Completion 2027-09-11 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | Up to the end of four cycles of treatment (1 cycle = 28 days)
  Will be defined as complete response, partial response, marrow complete response, or hematological improvement. Will be estimated for all patients along with the 95% confidence interval.
Incidence of adverse events | Up to 1 year
  The severity of the toxicities will be graded according to National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. The number and percent of subjects with treatment-emergent adverse events will be summarized according to intensity and drug relationship, and categorized by System Organ Class and preferred term by dose level/part. All reported adverse events that occur after signing informed consent will be included in the analysis of all reported adverse events. Exposure to study drug and reasons for discontinuation of study drug will be tabulated.

SECONDARY OUTCOMES:
Overall survival | Time from treatment start till death or last follow-up, assessed up to 1 year
  Will be listed and summarized by the Kaplan-Meier estimator, if needed.
Duration of response | Time from the first documented onset of partial response or complete response to the date of progressive disease/relapse, assessed up to 1 year
  Will be listed and summarized by the Kaplan-Meier estimator, if needed.
Leukemia free survival | Time from treatment start to transformation to acute myeloid leukemia or death, whichever comes first, assessed up to 1 year
  Will be listed and summarized by the Kaplan-Meier estimator, if needed.
Relapse-free survival | Time from start of response to the date of event defined as the first documented progressive disease/relapse or death, whichever comes first, assessed up to 1 year
  Will be listed and summarized by the Kaplan-Meier estimator, if needed.

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo M Bravo, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org